CLINICAL TRIAL: NCT01163799
Title: A Pilot Study to Assess the Safety and Efficacy of Alefacept in de Novo Kidney Transplant Recipients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Noted increased risks, greater than expected for standard of care therapy.
Sponsor: Northwestern University (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, M. Javeed Ansari, Assistant Professor of Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 00029396; 640 5442000 60026221 01 (Other: Northwestern University Internal Tracking Number)
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Transplant; Failure, Kidney
Keywords: Kidney; Transplant; Northwestern; Calcineurin Inhibitor; Corticosteroids; Steroid avoidance
MeSH Terms: interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alefacept (ASP0485) (Experimental): Safety and efficacy of alefacept in combination with alemtuzumab induction and calcineurin inhibitor (CNI) and corticosteroid withdrawal.
  Interventions: Drug: Alefacept (ASP0485)

INTERVENTIONS:
Drug: Alefacept (ASP0485) — Withdrawal of calcineurin inhibitor at 30 days post-transplant. Administer Alefacept 7.5 mg post-op day 0, post-op day 2 given IV; Alefacept 15 mg SQ X 12 weeks, then monthly until Month 12.
  Other Names: ASP0485

SUMMARY:
The purpose of this study is to assess Alefacept in combination with alemtuzumab induction and calcineurin inhibitor and corticosteroid withdrawal.

DETAILED DESCRIPTION:
This is a single center, investigator initiated, pilot study to assess the safety and efficacy of Alefacept in combination with Alemtuzumab induction and Myfortic with rapid steroid and calcineurin inhibitor withdrawal in de novo Kidney transplant recipients. Induction therapy involves single dose Alemtuzumab and steroids peri-operatively. Tacrolimus will be administered for the first 30 days post-transplantation. Alefacept will be administered IV for the first two doses followed by subcutaneous injections weekly until 12 weeks post-transplant followed by monthly injections for the rest of the duration of the study. The primary outcomes are safety and efficacy outcomes, including biopsy proven acute rejection episodes, infectious complications or other serious adverse events. Secondary outcomes include T-helper differentiation, cytokine production and T regulatory cell generation assessed by immune monitoring assays.

ELIGIBILITY:
Inclusion Criteria:

* Institutional Review Board (IRB) approved written Informed Consent and Health Insurance Portability and Accountability Act (HIPAA) Authorization for U.S. sites, or equivalent privacy language as per national regulations, obtained from the subject or legally authorized representative prior to study-related procedures (including withdrawal of prohibited medication, if applicable)
* Recipient of a kidney from a non-HLA identical related living donor, a non- related living donor, or deceased donor
* Recipient of a de novo kidney transplant
* ≥ 18 years of age
* Anticipated to receive first oral dose of tacrolimus within 48 hours of transplant procedure
* Female subjects of child bearing potential must have a negative urine or serum pregnancy test, and must agree to maintain effective birth control during the study

Healthy donor is eligible for the blood draw if:

* Institutional Review Board (IRB) approved written Informed Consent and Health Insurance Portability and Accountability Act (HIPAA) Authorization for U.S. sites, or equivalent privacy language as per national regulations, is obtained from subject prior to any study-related procedures
* Subject is a donor to a de novo kidney transplant subject who is enrolled in the study or a self declared healthy volunteer who is not a kidney donor for a subject enrolled in the study
* ≥ 18 years of age

Exclusion Criteria:

* Previously received or is receiving an organ transplant other than a kidney
* Sensitivity to iodine
* Will receive a transplant from a non-heart beating donor (donation after cardiac death - DCD)
* Receives a transplant from an HLA identical related living donor
* Will receive a solitary kidney from a deceased donor < 5 years of age
* Will receive a kidney with an anticipated cold ischemia time (CIT) of > 30 hours
* Will receive an ABO incompatible donor kidney
* Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV)
* Recipient has a positive T or B cell crossmatch by investigational site's standard method of determination. For recipients where a flow cytometry crossmatch is performed and is positive in either T or B cell testing, recipients are excluded only if donor specific, anti-HLA antibody is detected by flow cytometry based, specific anti-HLA antibody testing.
* Current malignancy or a history of malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully
* Significant liver disease
* Serologically negative for cytomegalovirus (CMV) with serologically positive CMV donor
* Serologically negative for Epstein Barr virus
* Has received intravenous immunoglobulin (IVIG) therapy in the three months prior to first dose of study drug
* Uncontrolled concomitant infection or any other unstable medical condition that could interfere with the study objectives
* Concurrently participating in another drug study or has received an investigational drug within 28 days prior to transplant
* Known hypersensitivity to alefacept, alemtuzumab, tacrolimus, mycophenolic acid, corticosteroids, or any of their components
* Any form of substance abuse, psychiatric disorder, or a condition that in the opinion of the Investigator could invalidate communication with the Investigator
* Subject is pregnant or lactating
* Subject is unlikely to comply with the visits scheduled in the protocol
* Subject will receive a kidney transplant from an expanded criteria donor (ECD)
* Will receive a kidney transplant from a CDC high risk donor

Healthy donor subject will be excluded from participation if any of the following apply:

* Unable to comprehend the investigational nature of the protocol participation
* Complete blood count results determined to be outside the normal ranges

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Incidence of first biopsy- proven acute rejection (Banff Grade≥ 1) (BCAR rate) and infections | At 12 months post-transplant
  To assess the safety and efficacy of alefacept in combination with a single dose of alemtuzamab induction and Enteric coated Mycophenolic sodium with calcineurin inhibitor withdrawal and rapid elimination of corticosteroids by examining the incidence of first biopsy-proven acute rejection (Banff Grade≥ 1) (BCAR rate) and the incidence and clinical presentation of infections.

SECONDARY OUTCOMES:
Affect on Immune cells | Up to 12 months post-transplant
  To assess how alefacept affects T-cell differentiation, memory, and immunoregulatory T-cell homeostasis, B-cells and cytokine/chemokine profile by using various immune monitoring assays.
Assess secondary outcome measures of efficacy and safety | Upto 12 months post-transplant
  At 12 months: Patient/graft survival rates, BCAR rate, Maximum grade of acute rejection with BCAR, Incidence of clinically-treated acute rejections, Incidence of anti-lymphocyte antibody therapy for treatment of rejection, Incidence of multiple rejection episodes, Incidence of treatment failure (defined as death, graft loss, biopsy-confirmed acute rejection, lost to follow-up or early discontinuation of treatment regimen), Incidence of leucopenia, Incidence of bacterial, fungal, viral, or parasitic infection. At 6 & 12 months: Serum creatinine, GFR by iohexol clearance. Time to first BCAR

CONTACTS AND LOCATIONS:
Overall Officials: M. Javeed Ansari, MD, Principal Investigator — Northwestern Universiy, Northwestern Memorial Hospital
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Ansari MJ, Sayegh MH. The arduous road to achieving an immunosuppression-free state in kidney transplant recipients. Nat Clin Pract Nephrol. 2007 Sep;3(9):464-5. doi: 10.1038/ncpneph0568. Epub 2007 Jul 24. No abstract available. PMID 17646858
- [Background] Antonysamy MA, Fanslow WC, Fu F, Li W, Qian S, Troutt AB, Thomson AW. Evidence for a role of IL-17 in alloimmunity: a novel IL-17 antagonist promotes heart graft survival. Transplant Proc. 1999 Feb-Mar;31(1-2):93. doi: 10.1016/s0041-1345(98)01453-5. No abstract available. PMID 10083023
- [Background] Beninga J, Kropff B, Mach M. Comparative analysis of fourteen individual human cytomegalovirus proteins for helper T cell response. J Gen Virol. 1995 Jan;76 ( Pt 1):153-60. doi: 10.1099/0022-1317-76-1-153. PMID 7844526
- [Background] Besse T, Malaise J, Mourad M, Pirson Y, Hope J, Awwad M, White-Scharf M, Squifflet JP. Prevention of rejection with BTI-322 after renal transplantation (results at 9 months). Transplant Proc. 1997 Aug;29(5):2425-6. doi: 10.1016/s0041-1345(97)00432-6. No abstract available. PMID 9270793
- [Background] Bishop DK, Chan Wood S, Eichwald EJ, Orosz CG. Immunobiology of allograft rejection in the absence of IFN-gamma: CD8+ effector cells develop independently of CD4+ cells and CD40-CD40 ligand interactions. J Immunol. 2001 Mar 1;166(5):3248-55. doi: 10.4049/jimmunol.166.5.3248. PMID 11207279
- [Background] Bobadilla JL, Love RB, Jankowska-Gan E, Xu Q, Haynes LD, Braun RK, Hayney MS, Munoz del Rio A, Meyer K, Greenspan DS, Torrealba J, Heidler KM, Cummings OW, Iwata T, Brand D, Presson R, Burlingham WJ, Wilkes DS. Th-17, monokines, collagen type V, and primary graft dysfunction in lung transplantation. Am J Respir Crit Care Med. 2008 Mar 15;177(6):660-8. doi: 10.1164/rccm.200612-1901OC. Epub 2008 Jan 3. PMID 18174545
- [Background] Burlingham WJ, Love RB, Jankowska-Gan E, Haynes LD, Xu Q, Bobadilla JL, Meyer KC, Hayney MS, Braun RK, Greenspan DS, Gopalakrishnan B, Cai J, Brand DD, Yoshida S, Cummings OW, Wilkes DS. IL-17-dependent cellular immunity to collagen type V predisposes to obliterative bronchiolitis in human lung transplants. J Clin Invest. 2007 Nov;117(11):3498-506. doi: 10.1172/JCI28031. PMID 17965778
- [Background] Chamian F, Lin SL, Lee E, Kikuchi T, Gilleaudeau P, Sullivan-Whalen M, Cardinale I, Khatcherian A, Novitskaya I, Wittkowski KM, Krueger JG, Lowes MA. Alefacept (anti-CD2) causes a selective reduction in circulating effector memory T cells (Tem) and relative preservation of central memory T cells (Tcm) in psoriasis. J Transl Med. 2007 Jun 7;5:27. doi: 10.1186/1479-5876-5-27. PMID 17555598
- [Background] Chisholm PL, Williams CA, Jones WE, Majeau GR, Oleson FB, Burrus-Fischer B, Meier W, Hochman PS. The effects of an immunomodulatory LFA3-IgG1 fusion protein on nonhuman primates. Ther Immunol. 1994 Aug;1(4):205-16. PMID 7584496
- [Background] Cooper JC, Morgan G, Harding S, Subramanyam M, Majeau GR, Moulder K, Alexander DR. Alefacept selectively promotes NK cell-mediated deletion of CD45R0+ human T cells. Eur J Immunol. 2003 Mar;33(3):666-75. doi: 10.1002/eji.200323586. PMID 12616487
- [Background] Crawford K, Gabuzda D, Pantazopoulos V, Xu J, Clement C, Reinherz E, Alper CA. Circulating CD2+ monocytes are dendritic cells. J Immunol. 1999 Dec 1;163(11):5920-8. PMID 10570278
- [Background] Crispim JC, Grespan R, Martelli-Palomino G, Rassi DM, Costa RS, Saber LT, Cunha FQ, Donadi EA. Interleukin-17 and kidney allograft outcome. Transplant Proc. 2009 Jun;41(5):1562-4. doi: 10.1016/j.transproceed.2009.01.092. PMID 19545679
- [Background] da Silva AJ, Brickelmaier M, Majeau GR, Li Z, Su L, Hsu YM, Hochman PS. Alefacept, an immunomodulatory recombinant LFA-3/IgG1 fusion protein, induces CD16 signaling and CD2/CD16-dependent apoptosis of CD2(+) cells. J Immunol. 2002 May 1;168(9):4462-71. doi: 10.4049/jimmunol.168.9.4462. PMID 11970990
- [Background] Dasgeb B, Holzman G, Phillips TJ. An extended 16-week course of alefacept in conjunction with reduced T-cell monitoring for the treatment of chronic plaque psoriasis. Poster P2720, American Academy of Dermatology 2005 Annual Meeting, New Orleans, Louisiana, February 2005.
- [Background] Dhanireddy KK, Bruno DA, Zhang X, Leopardi FV, Johnson LB, et al. Alefacept (LFA-3-Ig), portal venous donor specific transfusion, and sirolimus prolong renal allograft survival in non-human primates. Abstract 1627, American College of Surgeons 2006 Clinical Congress, Poster Session: Primate Models 2006 Jul 24.
- [Background] Di Pucchio T, Lapenta C, Santini SM, Logozzi M, Parlato S, Belardelli F. CD2+/CD14+ monocytes rapidly differentiate into CD83+ dendritic cells. Eur J Immunol. 2003 Feb;33(2):358-67. doi: 10.1002/immu.200310010. PMID 12548567
- [Background] Dustin ML, Springer TA. Role of lymphocyte adhesion receptors in transient interactions and cell locomotion. Annu Rev Immunol. 1991;9:27-66. doi: 10.1146/annurev.iy.09.040191.000331. PMID 1716919
- [Background] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697
- [Background] Ellis CN, Krueger GG; Alefacept Clinical Study Group. Treatment of chronic plaque psoriasis by selective targeting of memory effector T lymphocytes. N Engl J Med. 2001 Jul 26;345(4):248-55. doi: 10.1056/NEJM200107263450403. PMID 11474662
- [Background] Evans HG, Suddason T, Jackson I, Taams LS, Lord GM. Optimal induction of T helper 17 cells in humans requires T cell receptor ligation in the context of Toll-like receptor-activated monocytes. Proc Natl Acad Sci U S A. 2007 Oct 23;104(43):17034-9. doi: 10.1073/pnas.0708426104. Epub 2007 Oct 17. PMID 17942669
- [Background] Fabrega E, Lopez-Hoyos M, San Segundo D, Casafont F, Pons-Romero F. Changes in the serum levels of interleukin-17/interleukin-23 during acute rejection in liver transplantation. Liver Transpl. 2009 Jun;15(6):629-33. doi: 10.1002/lt.21724. PMID 19479806
- [Background] Gamadia LE, Remmerswaal EB, Weel JF, Bemelman F, van Lier RA, Ten Berge IJ. Primary immune responses to human CMV: a critical role for IFN-gamma-producing CD4+ T cells in protection against CMV disease. Blood. 2003 Apr 1;101(7):2686-92. doi: 10.1182/blood-2002-08-2502. Epub 2002 Oct 31. PMID 12411292
- [Background] Gandhi MK, Khanna R. Human cytomegalovirus: clinical aspects, immune regulation, and emerging treatments. Lancet Infect Dis. 2004 Dec;4(12):725-38. doi: 10.1016/S1473-3099(04)01202-2. PMID 15567122
- [Background] Gold MH, Hamilton TK, Rynearson A, Mathes B. An open-label community-based study of an extended course of alefacept in the treatment of chronic plaque psoriasis. Poster P2722, American Academy of Dermatology 2005 Annual Meeting, New Orleans, Louisiana, February 2005.
- [Background] Gonwa T, Mendez R, Yang HC, Weinstein S, Jensik S, Steinberg S; Prograf Study Group. Randomized trial of tacrolimus in combination with sirolimus or mycophenolate mofetil in kidney transplantation: results at 6 months. Transplantation. 2003 Apr 27;75(8):1213-20. doi: 10.1097/01.TP.0000062837.99400.60. PMID 12717205
- [Background] Gribetz CH, Blum R, Brady C, Cohen S, Lebwohl M. An extended 16-week course of alefacept in the treatment of chronic plaque psoriasis. J Am Acad Dermatol. 2005 Jul;53(1):73-5. doi: 10.1016/j.jaad.2005.03.053. PMID 15965424
- [Background] Humar A, Michaels M; AST ID Working Group on Infectious Disease Monitoring. American Society of Transplantation recommendations for screening, monitoring and reporting of infectious complications in immunosuppression trials in recipients of organ transplantation. Am J Transplant. 2006 Feb;6(2):262-74. doi: 10.1111/j.1600-6143.2005.01207.x. PMID 16426310
- [Background] Ibrahim S, Dawson DV, Sanfilippo F. Predominant infiltration of rejecting human renal allografts with T cells expressing CD8 and CD45RO. Transplantation. 1995 Mar 15;59(5):724-8. doi: 10.1097/00007890-199503150-00015. PMID 7886800
- [Background] Jeong H, Kaplan B. Therapeutic monitoring of mycophenolate mofetil. Clin J Am Soc Nephrol. 2007 Jan;2(1):184-91. doi: 10.2215/CJN.02860806. Epub 2006 Nov 8. No abstract available. PMID 17699403
- [Background] Johnson C, Ahsan N, Gonwa T, Halloran P, Stegall M, Hardy M, Metzger R, Shield C 3rd, Rocher L, Scandling J, Sorensen J, Mulloy L, Light J, Corwin C, Danovitch G, Wachs M, van Veldhuisen P, Salm K, Tolzman D, Fitzsimmons WE. Randomized trial of tacrolimus (Prograf) in combination with azathioprine or mycophenolate mofetil versus cyclosporine (Neoral) with mycophenolate mofetil after cadaveric kidney transplantation. Transplantation. 2000 Mar 15;69(5):834-41. doi: 10.1097/00007890-200003150-00028. PMID 10755536
- [Background] Jones ND, Van Maurik A, Hara M, Spriewald BM, Witzke O, Morris PJ, Wood KJ. CD40-CD40 ligand-independent activation of CD8+ T cells can trigger allograft rejection. J Immunol. 2000 Jul 15;165(2):1111-8. doi: 10.4049/jimmunol.165.2.1111. PMID 10878390
- [Background] Kaplon RJ, Hochman PS, Michler RE, Kwiatkowski PA, Edwards NM, Berger CL, Xu H, Meier W, Wallner BP, Chisholm P, Marboe CC. Short course single agent therapy with an LFA-3-IgG1 fusion protein prolongs primate cardiac allograft survival. Transplantation. 1996 Feb 15;61(3):356-63. doi: 10.1097/00007890-199602150-00004. PMID 8610340
- [Background] Kondo T, Takata H, Matsuki F, Takiguchi M. Cutting edge: Phenotypic characterization and differentiation of human CD8+ T cells producing IL-17. J Immunol. 2009 Feb 15;182(4):1794-8. doi: 10.4049/jimmunol.0801347. PMID 19201830
- [Background] Krueger GG, Papp KA, Stough DB, Loven KH, Gulliver WP, Ellis CN; Alefacept Clinical Study Group. A randomized, double-blind, placebo-controlled phase III study evaluating efficacy and tolerability of 2 courses of alefacept in patients with chronic plaque psoriasis. J Am Acad Dermatol. 2002 Dec;47(6):821-33. doi: 10.1067/mjd.2002.127247. PMID 12451365
- [Background] Lerut J, Van Thuyne V, Mathijs J, Lemaire J, Talpe S, Roggen F, Ciccarelli O, Zuckermann M, Goffette P, Hope J, Gianello P, Bazin H, Cornet A, Rahier J, Latinne D. Anti-CD2 monoclonal antibody and tacrolimus in adult liver transplantation. Transplantation. 2005 Nov 15;80(9):1186-93. doi: 10.1097/01.tp.0000173996.81192.f9. PMID 16314784
- [Background] Loong CC, Hsieh HG, Lui WY, Chen A, Lin CY. Evidence for the early involvement of interleukin 17 in human and experimental renal allograft rejection. J Pathol. 2002 Jul;197(3):322-32. doi: 10.1002/path.1117. PMID 12115878 (Retraction: PMID 23130366 J Pathol. 2012 Oct;228(2):260)
- [Background] Majeau GR, Meier W, Jimmo B, Kioussis D, Hochman PS. Mechanism of lymphocyte function-associated molecule 3-Ig fusion proteins inhibition of T cell responses. Structure/function analysis in vitro and in human CD2 transgenic mice. J Immunol. 1994 Mar 15;152(6):2753-67. PMID 7511625
- [Background] Mendez R, Gonwa T, Yang HC, Weinstein S, Jensik S, Steinberg S; Prograf Study Group. A prospective, randomized trial of tacrolimus in combination with sirolimus or mycophenolate mofetil in kidney transplantation: results at 1 year. Transplantation. 2005 Aug 15;80(3):303-9. doi: 10.1097/01.tp.0000167757.63922.42. PMID 16082323
- [Background] Miller GT, Hochman PS, Meier W, Tizard R, Bixler SA, Rosa MD, Wallner BP. Specific interaction of lymphocyte function-associated antigen 3 with CD2 can inhibit T cell responses. J Exp Med. 1993 Jul 1;178(1):211-22. doi: 10.1084/jem.178.1.211. PMID 7686212
- [Background] Miller J, Mendez R, Pirsch JD, Jensik SC. Safety and efficacy of tacrolimus in combination with mycophenolate mofetil (MMF) in cadaveric renal transplant recipients. FK506/MMF Dose-Ranging Kidney Transplant Study Group. Transplantation. 2000 Mar 15;69(5):875-80. doi: 10.1097/00007890-200003150-00035. PMID 10755543
- [Background] Mourad M, Besse T, Malaise J, Baldi A, Latinne D, Bazin H, Pirson Y, Hope J, Squifflet JP. BTI-322 for acute rejection after renal transplantation. Transplant Proc. 1997 Aug;29(5):2353. doi: 10.1016/s0041-1345(97)00398-9. No abstract available. PMID 9270759
- [Background] Newell KA, He G, Guo Z, Kim O, Szot GL, Rulifson I, Zhou P, Hart J, Thistlethwaite JR, Bluestone JA. Cutting edge: blockade of the CD28/B7 costimulatory pathway inhibits intestinal allograft rejection mediated by CD4+ but not CD8+ T cells. J Immunol. 1999 Sep 1;163(5):2358-62. PMID 10452966
- [Background] Olson DP, Dombkowski DM, Kelliher AS, Pontillo C, Anderson DC, Preffer FI. Differential expression of cell surface antigens on subsets of CD4+ and CD8+ T cells. Med Sci Monit. 2004 Sep;10(9):BR339-45. Epub 2004 Aug 20. PMID 15328479
- [Background] Park H, Li Z, Yang XO, Chang SH, Nurieva R, Wang YH, Wang Y, Hood L, Zhu Z, Tian Q, Dong C. A distinct lineage of CD4 T cells regulates tissue inflammation by producing interleukin 17. Nat Immunol. 2005 Nov;6(11):1133-41. doi: 10.1038/ni1261. Epub 2005 Oct 2. PMID 16200068
- [Background] Preston EH, Xu H, Dhanireddy KK, Pearl JP, Leopardi FV, Starost MF, Hale DA, Kirk AD. IDEC-131 (anti-CD154), sirolimus and donor-specific transfusion facilitate operational tolerance in non-human primates. Am J Transplant. 2005 May;5(5):1032-41. doi: 10.1111/j.1600-6143.2005.00796.x. PMID 15816883
- [Background] Putnam Associates, from the results of a survey (funded by Astellas Pharma US, Inc.) conducted at the 2004 American Transplant Congress July 14, 2004.
- [Background] Valujskikh A, Pantenburg B, Heeger PS. Primed allospecific T cells prevent the effects of costimulatory blockade on prolonged cardiac allograft survival in mice. Am J Transplant. 2002 Jul;2(6):501-9. doi: 10.1034/j.1600-6143.2002.20603.x. PMID 12118893
- [Background] Van Kooten C, Boonstra JG, Paape ME, Fossiez F, Banchereau J, Lebecque S, Bruijn JA, De Fijter JW, Van Es LA, Daha MR. Interleukin-17 activates human renal epithelial cells in vitro and is expressed during renal allograft rejection. J Am Soc Nephrol. 1998 Aug;9(8):1526-34. doi: 10.1681/ASN.V981526. PMID 9697677
- [Background] Vanaudenaerde BM, Dupont LJ, Wuyts WA, Verbeken EK, Meyts I, Bullens DM, Dilissen E, Luyts L, Van Raemdonck DE, Verleden GM. The role of interleukin-17 during acute rejection after lung transplantation. Eur Respir J. 2006 Apr;27(4):779-87. doi: 10.1183/09031936.06.00019405. PMID 16585086
- [Background] Sester M, Sester U, Gartner BC, Girndt M, Meyerhans A, Kohler H. Dominance of virus-specific CD8 T cells in human primary cytomegalovirus infection. J Am Soc Nephrol. 2002 Oct;13(10):2577-84. doi: 10.1097/01.asn.0000030141.41726.52. PMID 12239248
- [Background] Sester M, Sester U, Gartner B, Heine G, Girndt M, Mueller-Lantzsch N, Meyerhans A, Kohler H. Levels of virus-specific CD4 T cells correlate with cytomegalovirus control and predict virus-induced disease after renal transplantation. Transplantation. 2001 May 15;71(9):1287-94. doi: 10.1097/00007890-200105150-00018. PMID 11397964
- [Background] Solez K, Colvin RB, Racusen LC, Sis B, Halloran PF, Birk PE, Campbell PM, Cascalho M, Collins AB, Demetris AJ, Drachenberg CB, Gibson IW, Grimm PC, Haas M, Lerut E, Liapis H, Mannon RB, Marcus PB, Mengel M, Mihatsch MJ, Nankivell BJ, Nickeleit V, Papadimitriou JC, Platt JL, Randhawa P, Roberts I, Salinas-Madriga L, Salomon DR, Seron D, Sheaff M, Weening JJ. Banff '05 Meeting Report: differential diagnosis of chronic allograft injury and elimination of chronic allograft nephropathy ('CAN'). Am J Transplant. 2007 Mar;7(3):518-26. doi: 10.1111/j.1600-6143.2006.01688.x. PMID 17352710
- [Background] Squifflet JP, Backman L, Claesson K, Dietl KH, Ekberg H, Forsythe JL, Kunzendorf U, Heemann U, Land W, Morales JM, Muhlbacher F, Talbot D, Taube D, Tyden G, van Hooff J, Schleibner S, Vanrenterghem Y; European Tacrolimus-MMF Renal Study Group. Dose optimization of mycophenolate mofetil when administered with a low dose of tacrolimus in cadaveric renal transplant recipients. Transplantation. 2001 Jul 15;72(1):63-9. doi: 10.1097/00007890-200107150-00014. PMID 11468536
- [Background] Squifflet JP, Besse T, Malaise J, Mourad M, Delcorde C, Hope JA, Pirson Y. BTI-322 for induction therapy after renal transplantation: a randomized study. Transplant Proc. 1997 Feb-Mar;29(1-2):317-9. doi: 10.1016/s0041-1345(96)00282-5. No abstract available. PMID 9123018
- [Background] Sultan P, Schechner JS, McNiff JM, Hochman PS, Hughes CC, Lorber MI, Askenase PW, Pober JS. Blockade of CD2-LFA-3 interactions protects human skin allografts in immunodeficient mouse/human chimeras. Nat Biotechnol. 1997 Aug;15(8):759-62. doi: 10.1038/nbt0897-759. PMID 9255790
- [Background] Walter EA, Greenberg PD, Gilbert MJ, Finch RJ, Watanabe KS, Thomas ED, Riddell SR. Reconstitution of cellular immunity against cytomegalovirus in recipients of allogeneic bone marrow by transfer of T-cell clones from the donor. N Engl J Med. 1995 Oct 19;333(16):1038-44. doi: 10.1056/NEJM199510193331603. PMID 7675046
- [Background] Wu Z, Bensinger SJ, Zhang J, Chen C, Yuan X, Huang X, Markmann JF, Kassaee A, Rosengard BR, Hancock WW, Sayegh MH, Turka LA. Homeostatic proliferation is a barrier to transplantation tolerance. Nat Med. 2004 Jan;10(1):87-92. doi: 10.1038/nm965. Epub 2003 Nov 30. PMID 14647496
- [Background] Yuan X, Ansari MJ, D'Addio F, Paez-Cortez J, Schmitt I, Donnarumma M, Boenisch O, Zhao X, Popoola J, Clarkson MR, Yagita H, Akiba H, Freeman GJ, Iacomini J, Turka LA, Glimcher LH, Sayegh MH. Targeting Tim-1 to overcome resistance to transplantation tolerance mediated by CD8 T17 cells. Proc Natl Acad Sci U S A. 2009 Jun 30;106(26):10734-9. doi: 10.1073/pnas.0812538106. Epub 2009 Jun 15. PMID 19528638
- [Background] Yuan X, Paez-Cortez J, Schmitt-Knosalla I, D'Addio F, Mfarrej B, Donnarumma M, Habicht A, Clarkson MR, Iacomini J, Glimcher LH, Sayegh MH, Ansari MJ. A novel role of CD4 Th17 cells in mediating cardiac allograft rejection and vasculopathy. J Exp Med. 2008 Dec 22;205(13):3133-44. doi: 10.1084/jem.20081937. Epub 2008 Dec 1. PMID 19047438
- [Background] Zhai Y, Meng L, Gao F, Busuttil RW, Kupiec-Weglinski JW. Allograft rejection by primed/memory CD8+ T cells is CD154 blockade resistant: therapeutic implications for sensitized transplant recipients. J Immunol. 2002 Oct 15;169(8):4667-73. doi: 10.4049/jimmunol.169.8.4667. PMID 12370407